CLINICAL TRIAL: NCT03717155
Title: A Phase IIa, Single-arm, Multicenter Study to Investigate the Clinical Activity and Safety of Avelumab in Combination With Cetuximab Plus Gemcitabine and Cisplatin in Participants With Advanced Squamous NSCLC
Brief Title: Study of Avelumab and Cetuximab Plus Gemcitabine and Cisplatin in Participants With NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS201944_0170; 2018-001529-24 (EudraCT Number)
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Results first posted 2021-11-09 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-04

CONDITIONS: Squamous Non-Small Cell Lung Cancer
Keywords: Avelumab; Cetuximab; Cisplatin; Gemcitabine; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — avelumab; Cetuximab; Gemcitabine; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avelumab and Cetuximab (Experimental): Participants received 800 milligrams Avelumab, 1250 milligrams per square meter (mg/m^2) gemcitabine on Day 1 and Day 8, cisplatin at a dose of 75 mg/m^2 on Day 1 along with 250 mg/m2 body surface area Cetuximab on Day 1 and 500 mg/m2 body surface area on Day 8 of each cycle as intravenous (IV) infusions up to maximum of 4 cycles (each cycle is of 3 weeks) until disease progression or unacceptable toxicities. In case of cisplatin toxicities, participants were switched to carboplatin at a dose of target area under the serum concentration-time curve of 5 (AUC 5) on Day 1 for the remainder of cycles. Subsequently participants were administered with avelumab and cetuximab as IV infusion at the dose of 800 mg and 500 mg/m^2 respectively, every 2 weeks in the Maintenance phase until disease progression or unacceptable toxicities.
  Interventions: Drug: Avelumab; Drug: Cetuximab; Drug: Gemcitabine; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: Avelumab — Participants received avelumab intravenous infusions at a dose of 800 milligram (mg) on Day 1 and Day 8 of each 3-week cycle for the first 4 cycles. Thereafter, administered every 2 weeks in the Maintenance phase until disease progression or unacceptable toxicities.
Drug: Cetuximab — Participants received cetuximab intravenous infusions at a dose of 250 milligram per meter square (mg/m^2) body surface area on Day 1 and 500 mg/m^2 body surface area on Day 8 of first 4 cycles of concurrent chemotherapy. Thereafter, administered given at a dose of 500 mg/m^2 intravenous every 2 weeks in the Maintenance phase, until disease progression or unacceptable toxicities.
Drug: Gemcitabine — Participants received gemcitabine intravenous infusions at a dose of 1250 mg/m^2 body surface area on Day 1 and Day 8 in 3-week cycles up to a maximum of 4 cycles, until disease progression or unacceptable toxicities.
Drug: Cisplatin — Participants received cisplatin intravenous infusions at a dose of 75 mg/m^2 body surface area on Day 1 of 3-week cycles up to a maximum of 4 cycles, until disease progression or unacceptable toxicities.
Drug: Carboplatin — In case of cisplatin toxicities, participants were switched to carboplatin at a dose of target area under the serum concentration-time curve of 5 (AUC 5) on Day 1 for the remainder of cycles.

SUMMARY:
The main purpose of the study was to investigate the clinical activity and safety of avelumab in combination with cetuximab plus gemcitabine and cisplatin in participants with treatment-naïve advanced squamous non-small-cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed Stage IV metastatic or recurrent (Stage IV) NSCLC of squamous histology
* Availability of formalin-fixed paraffin-embedded (FFPE) block containing tumor tissue or a minimum of 15 (preferably 25) unstained tumor slides (cut within 1 week) suitable for Programmed death ligand 1 (PD-L1) expression and epidermal growth factor receptor (EGFR) expression/amplification assessments
* At least 1 measurable lesion per response evaluation criteria in solid tumors (RECIST) v1.1 criteria
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1 at study entry
* Adequate hematological, hepatic and renal function
* Estimated life expectancy of at least 3 months
* Can give signed informed consent
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants whose tumor disease harbors an activating EGFR mutation or ALK rearrangement. Participants with tumors of unknown EGFR or ALK status will require testing only in never smokers
* All participants with brain metastases with protocol defined exceptions
* Previous malignant disease (other than NSCLC) within the last 5 years (except adequately treated non-melanoma skin cancers, carcinoma in situ of skin, bladder, cervix, colon/rectum, breast, or prostate) unless a complete remission without further recurrence was achieved at least 2 years prior to study entry and the participant was deemed to have been cured with no additional therapy required or anticipated to be required
* Active infection requiring systemic therapy
* Known history of human immunodeficiency virus or known acquired immunodeficiency syndrome
* Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV ribonucleic acid (RNA) if anti-HCV antibody screening test positive)
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent
* Interstitial parenchymal lung disease
* Pregnancy or lactation
* Known alcohol or drug abuse as determined by the Investigator
* History of uncontrolled intercurrent illness
* Clinically significant (that is active) cardiovascular disease
* Known history of inflammatory colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis
* Any psychiatric condition that would prohibit the understanding or rendering of informed consent or that would limit compliance with study requirements
* Prior/Concomitant Therapy as described in protocol
* Use of any investigational drug within 28 days before the start of study treatment
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (20):
- Hungary (6):
  - Semmelweis Egyetem - Pulmonologiai Klinika, Budapest
  - Debreceni Egyetem - Tudogyogyaszati Klinika, Debrecen
  - Petz Aladar Megyei Oktato Korhaz - Pulmonologiai Osztaly, Győr
  - Markusovszky Egyetemi Oktatokorhaz, Szombathely
  - Tudogyogyintezet Torokbalint - Onkopulmonologiai es Jarobeteg centrum, Törökbálint
  - Zala Megyei Szent Rafael Korhaz, Zalaegerszeg
- Serbia (3):
  - Clinical Center "Bezanijska kosa" - Department of Oncology, Belgrade
  - Clinical Center Kragujevac (no dept.), Belgrade
  - Institute for Pulmonary Diseases of Vojvodina, Kamenitz
- Spain (11):
  - Complejo Hospitalario Universitario A Coruña - Servicio de Oncologia, A Coruña
  - Hospital Universitari Quiron Dexeus - Servicio de Oncologia Medica, Barcelona
  - Hospital Universitari Vall d'Hebron - Dept of Oncology, Barcelona
  - Hospital General Universitario Gregorio Marañon - Servicio de Oncologia Medica, Madrid
  - Hospital Universitario 12 de Octubre - Servicio de Oncologia, Madrid
  - Hospital Universitario HM Madrid Sanchinarro - Servicio de Oncologia, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Virgen Macarena - Servicio de Oncologia, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe - Servicio de Oncologia Medica, Valencia
  - Hospital Clinico Universitario Lozano Blesa - Dept of Oncology, Zaragoza

REFERENCES:
- [Derived] Andric Z, Galffy G, Cobo Dols M, Szima B, Stojanovic G, Petrovic M, Felip E, Vicente Baz D, Ponce Aix S, Juan-Vidal O, Szalai Z, Losonczy G, Calles Blanco A, Bernabe R, Garcia Ledo G, Aguilar Hernandez A, Duecker K, Zhou D, Schroeder A, Guezel G, Ciardiello F. Avelumab in Combination With Cetuximab and Chemotherapy as First-Line Treatment for Patients With Advanced Squamous NSCLC. JTO Clin Res Rep. 2023 Jan 2;4(2):100461. doi: 10.1016/j.jtocrr.2022.100461. eCollection 2023 Feb. PMID 36718142
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS201944_0170
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 43 participants were enrolled in this study at different sites in Hungary, Serbia and Spain.
Period: Overall Study
Arm/Group | Avelumab and Cetuximab
Started | 43
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Avelumab and Cetuximab
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 43
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Confirmed Best Objective Response (BOR) According to Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1 Assessed by Investigator
Description: Confirmed BOR was defined as the percentage of participants who achieved confirmed complete responses (CR) or partial response (PR), according to RECIST version 1.1 assessed by the Investigator.CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30 percent (%) reduction from baseline in the sum of the longest diameter (SLD) of all lesions. Stable disease (SD)= Neither sufficient increase to qualify for progression of disease (PD) nor sufficient shrinkage to qualify for PR. PD: At least a 20 % increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. Confirmed CR=as at least two determinations of CR at least 4 weeks apart with no PD. Confirmed PR=as at least 2 determinations of PR or better (PR followed by PR or PR followed by CR), at least 4 weeks apart (not qualifying for a CR) with no PD in between. Percentage of Participants with confirmed BOR were reported.
Time Frame: Time from the first dose of study drug until occurrence of PD, death due to any cause (assessed up to 612 days)
Population: Full analysis set includes all participants who received at least one non-zero dose of any study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Avelumab and Cetuximab
Number analyzed (Participants) | 43
percentage of participants | 34.9 [21.0 to 50.9]

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Related Adverse Events (AEs), Treatment-Related Grade >=3 TEAEs and Immune-related Treatment Emergent AEs (irTEAEs)
Description: Adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug.Serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAE is defined as AEs starting or worsening after the first intake of the study drug. TEAEs include both Serious and non-serious TEAEs. irAEs included AEs that matches a preferred term on the list of pre-selected MedDRA terms. AEs with relationship to study treatment are reported as Treatment-related AEs. Treatment related AEs with grade 3 or more is also reported.
Time Frame: Time from the first dose of study drug assessed up to (941 days)
Population: Safety analysis set included all participants who received at least one non-zero dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab and Cetuximab
Number analyzed (Participants) | 43
Participants
  TEAEs | 41
  Treatment-Related AEs | 38
  Treatment Related Grade>=3 TEAEs | 24
  irTEAEs | 13

3. Secondary Outcome: Progression-Free Survival (PFS) Time Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Description: Progression free survival (PFS) is defined as the time (in months) from first treatment day to the date of the first documentation of objective progression of disease (PD) according to RECIST version 1.1 assessed by Investigator, or death due to any cause, whichever occurs first. PD is defined as at least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: Time from the first dose of study drug until occurrence of PD, death due to any cause (assessed up to 737 days)
Population: Full analysis set includes all participants who received at least one non-zero dose of any study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Avelumab and Cetuximab
Number analyzed (Participants) | 43
Months | 6.1 [4.3 to 9.0]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined for participants with confirmed complete response (CR) or partial response (PR), as the time from first documentation of confirmed response to the date of first documentation of progression of disease (PD) according to RECIST version 1.1 (assessed by Investigator) or death due to any cause or tumor assessment. Duration of objective response was assessed using Kaplan-Meier analysis. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the SLD of all lesions. PD: At least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: Time from the first dose of study drug until occurrence of PD, death due to any cause or last tumor assessment (assessed up to 612 days)
Population: Full analysis set included all participants who receive at least one non-zero dose of any study treatment. Here "Overall number of participants analyzed" signifies those participants who had confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Avelumab and Cetuximab
Number analyzed (Participants) | 15
Months | 7.1 [4.2 to 12.5]

5. Secondary Outcome: Immediate Observed Serum Concentration at End of Infusion (Ceoi) of Avelumab
Description: Ceoi is the serum concentration observed immediately at the end of infusion. This was taken directly from the observed Avelumab concentration-time data.
Time Frame: Pre-dose, 2 hours after end of infusion on Day 1, 8, 22 and 29; Pre-dose, 30 minutes after the end of infusion on Day 43, 50, 64, 71; Pre-dose, 3 hours after end of infusion on Day 85, 99, 113, 127, 169, 253, and 337
Population: Pharmacokinetic (PK) analysis set included all participants who receive at least one dose of avelumab and/or cetuximab, have no important events affecting PK, and provide at least one measurable post-dose concentration. Number of Participants Analyzed=participants evaluable for this outcome and Number analyzed=participants evaluated at specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Avelumab and Cetuximab
Number analyzed (Participants) | 40
microgram per milliliter (mcg/mL)
  Day 1 | 206 (26.6)
  Day 8: number analyzed (Participants) | 36
  Day 8 | 243 (23.8)
  Day 22: number analyzed (Participants) | 29
  Day 22 | 234 (24.1)
  Day 29: number analyzed (Participants) | 31
  Day 29 | 282 (26.8)
  Day 43: number analyzed (Participants) | 22
  Day 43 | 237 (30.5)
  Day 50: number analyzed (Participants) | 32
  Day 50 | 259 (38.9)
  Day 64: number analyzed (Participants) | 22
  Day 64 | 214 (67.6)
  Day 71: number analyzed (Participants) | 28
  Day 71 | 244 (43.8)
  Day 85: number analyzed (Participants) | 25
  Day 85 | 223 (33.3)
  Day 99: number analyzed (Participants) | 25
  Day 99 | 202 (62.4)
  Day 113: number analyzed (Participants) | 27
  Day 113 | 234 (29.7)
  Day 127: number analyzed (Participants) | 20
  Day 127 | 222 (55.1)
  Day 169: number analyzed (Participants) | 21
  Day 169 | 245 (20.8)
  Day 253: number analyzed (Participants) | 10
  Day 253 | 249 (28.7)
  Day 337: number analyzed (Participants) | 9
  Day 337 | 246 (38.6)

6. Secondary Outcome: Immediate Observed Serum Concentration at End of Infusion (Ceoi) of Cetuximab
Description: Ceoi is the serum concentration observed immediately at the end of infusion. This was taken directly from the observed cetuximab concentration-time data.
Time Frame: as for outcome 5
Population: PK analysis set included all participants who receive at least one dose of avelumab and/or cetuximab, have no important events affecting PK, and provide at least one measurable post-dose concentration. Number analyzed=participants evaluated at specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Avelumab and Cetuximab
Number analyzed (Participants) | 43
mcg/mL
  Day 1 | 109 (50.7)
  Day 8: number analyzed (Participants) | 35
  Day 8 | 198 (86.6)
  Day 22: number analyzed (Participants) | 28
  Day 22 | 124 (54.4)
  Day 29: number analyzed (Participants) | 30
  Day 29 | 260 (25.0)
  Day 43: number analyzed (Participants) | 22
  Day 43 | 154 (32.7)
  Day 50: number analyzed (Participants) | 30
  Day 50 | 238 (28.9)
  Day 64: number analyzed (Participants) | 21
  Day 64 | 159 (36.1)
  Day 71: number analyzed (Participants) | 27
  Day 71 | 262 (25.1)
  Day 85: number analyzed (Participants) | 25
  Day 85 | 239 (38.4)
  Day 99: number analyzed (Participants) | 25
  Day 99 | 252 (21.1)
  Day 113: number analyzed (Participants) | 26
  Day 113 | 250 (20.4)
  Day 127: number analyzed (Participants) | 21
  Day 127 | 245 (55.8)
  Day 169: number analyzed (Participants) | 20
  Day 169 | 297 (29.2)
  Day 253: number analyzed (Participants) | 10
  Day 253 | 269 (34.4)
  Day 337: number analyzed (Participants) | 9
  Day 337 | 304 (37.3)

7. Secondary Outcome: Serum Trough Concentration Levels (Ctrough) of Avelumab
Description: Ctrough is the serum concentration observed immediately before next dosing.
Time Frame: Pre-dose: Day 8, Day 22, Day 29, Day 43, Day 50, Day 64, Day 71, Day 85, Day 99, Day 113, Day 127, Day 169, Day 253 and Day 337
Population: PK analysis set included all participants who receive at least one dose of avelumab and/or cetuximab, have no important events affecting PK, and provide at least one measurable post-dose concentration. Number of Participants Analyzed=participants evaluable for this outcome and Number analyzed=participants evaluated at specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Avelumab and Cetuximab
Number analyzed (Participants) | 35
mcg/mL
  Day 8 | 28.8 (82.7)
  Day 22: number analyzed (Participants) | 29
  Day 22 | 13.6 (97.1)
  Day 29: number analyzed (Participants) | 31
  Day 29 | 42.4 (147.8)
  Day 43: number analyzed (Participants) | 22
  Day 43 | 15.6 (115.1)
  Day 50: number analyzed (Participants) | 32
  Day 50 | 56.4 (77.9)
  Day 64: number analyzed (Participants) | 22
  Day 64 | 19.7 (145.7)
  Day 71: number analyzed (Participants) | 27
  Day 71 | 58.2 (62.5)
  Day 85: number analyzed (Participants) | 25
  Day 85 | 21.5 (70.9)
  Day 99: number analyzed (Participants) | 25
  Day 99 | 21.2 (75.4)
  Day 113: number analyzed (Participants) | 27
  Day 113 | 19.4 (78.5)
  Day 127: number analyzed (Participants) | 21
  Day 127 | 18.1 (107.6)
  Day 169: number analyzed (Participants) | 21
  Day 169 | 19.3 (67.2)
  Day 253: number analyzed (Participants) | 10
  Day 253 | 17.0 (80.1)
  Day 337: number analyzed (Participants) | 9
  Day 337 | 20.8 (55.9)

8. Secondary Outcome: Serum Trough Concentration Levels (Ctrough) of Cetuximab
Description: Ctrough is the serum concentration observed immediately before next dosing.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Avelumab and Cetuximab
Number analyzed (Participants) | 32
mcg/mL
  Day 8 | 12.1 (90.0)
  Day 22: number analyzed (Participants) | 26
  Day 22 | 12.8 (63.7)
  Day 29: number analyzed (Participants) | 29
  Day 29 | 22.8 (73.3)
  Day 43: number analyzed (Participants) | 20
  Day 43 | 25.6 (103.7)
  Day 50: number analyzed (Participants) | 30
  Day 50 | 23.9 (118.1)
  Day 64: number analyzed (Participants) | 20
  Day 64 | 17.2 (157.9)
  Day 71: number analyzed (Participants) | 27
  Day 71 | 35.4 (110.4)
  Day 85: number analyzed (Participants) | 22
  Day 85 | 26.5 (119.4)
  Day 99: number analyzed (Participants) | 22
  Day 99 | 22.6 (117.3)
  Day 113: number analyzed (Participants) | 23
  Day 113 | 35.0 (59.0)
  Day 127: number analyzed (Participants) | 18
  Day 127 | 38.0 (63.6)
  Day 169: number analyzed (Participants) | 19
  Day 169 | 40.4 (62.2)
  Day 253: number analyzed (Participants) | 10
  Day 253 | 31.9 (237.7)
  Day 337: number analyzed (Participants) | 9
  Day 337 | 28.9 (204.9)

9. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the first treatment day to the date of death due to any cause. Overall survival was assessed using Kaplan-Meier analysis.
Time Frame: Time from the first dose of study drug until occurrence of death due to any cause (assessed up to 941 days)
Population: Full analysis set includes all participants who received at least one non-zero dose of any study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Avelumab and Cetuximab
Number analyzed (Participants) | 43
Months | 10.1 [8.6 to 14.5]

10. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody (ADA) of Avelumab
Description: The detection of antibodies to avelumab was performed using a validated immunoassay method with tiered testing of screening, confirmatory and titration. Number of participants with positive anti-drug antibody (ADA) of avelumab were reported.
Time Frame: Pre-dose up to 149 days
Population: ADA analysis set included all participants who received at least 1 dose of avelumab and/or cetuximab and have at least 1 valid ADA result.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab and Cetuximab
Number analyzed (Participants) | 43
Participants | 7

11. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody (ADA) of Cetuximab
Description: The detection of antibodies to cetuximab was performed using a validated immunoassay method with tiered testing of screening, confirmatory and titration. Number of participants with positive anti-drug antibody (ADA) of cetuximab were reported.
Time Frame: Pre-dose up to 149 days
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab and Cetuximab
Number analyzed (Participants) | 43
Participants | 1

ADVERSE EVENTS:
Time Frame: Time from the first dose of study drug until 941 days.
Arm/Group | Avelumab and Cetuximab
All-Cause Mortality (participants affected / at risk) | 30/43
Serious Adverse Events (participants affected / at risk) | 20/43
Other Adverse Events (participants affected / at risk) | 39/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab and Cetuximab (N=43)
Anaemia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Death (General disorders) | 1
Disease progression (General disorders) | 4
Non-cardiac chest pain (General disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Blood creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Seizure (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Dry gangrene (Vascular disorders) | 1
Femoral artery embolism (Vascular disorders) | 1
Peripheral artery thrombosis (Vascular disorders) | 1
Tachycardia (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab and Cetuximab (N=43)
Anaemia (Blood and lymphatic system disorders) | 19
Leukopenia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 7
Asthenia (General disorders) | 12
Fatigue (General disorders) | 7
Oedema peripheral (General disorders) | 3
Pyrexia (General disorders) | 6
Nasopharyngitis (Infections and infestations) | 3
Respiratory tract infection (Infections and infestations) | 3
Alanine aminotransferase increased (Investigations) | 6
Amylase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 4
Blood creatinine increased (Investigations) | 5
Neutrophil count decreased (Investigations) | 3
Transaminases increased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 16
Hyponatraemia (Metabolism and nutrition disorders) | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 22
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-08-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT03717155/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT03717155/SAP_001.pdf